CLINICAL TRIAL: NCT05597202
Title: Does the Hematopoietic Stem Cell Govern Residual Inflammatory Cardiovascular Risk in Type 2 Diabetes
Acronym: DOTAFLAME
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Dutch Heart Foundation (Other)
Responsible Party: Principal Investigator, Nordin Hanssen, Principal investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL80519.018.22
Record Dates: First submitted 2022-10-14; First posted 2022-10-27 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Type 2 Diabetes
Keywords: diabetes mellitus; dotatate; bone marrow; semaglutide; vascular inflammation; glp1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Will receive semaglutide treatment for 6 months, at the highest tolerable dose, up to a maximum of 2.0mg weekly.
  Interventions: Drug: Semaglutide, 2.0 mg/mL

INTERVENTIONS:
Drug: Semaglutide, 2.0 mg/mL — Semaglutide 2.0 mg/mL, administered subcutaneously once per week for a period of 6 months.

SUMMARY:
To study the effect of type 2 diabetes (T2D) on vascular wall inflammation and hematopoietic stem cell composition in vivo, and whether these changes can be reversed with glucagon like peptide 1 receptor (GLP1R)-agonism.

DETAILED DESCRIPTION:
We will use 68Ga-Dotatate PET/CT scans, bone marrow aspirations and peripheral blood analyses to determine the effect of type 2 diabetes on vascular wall inflammation, and hematopoietic stem cell composition, and whether these changes can be reversed using high dose semaglutide treatment, up to 2.0mg subcutaneously per week, for a period of six months.

ELIGIBILITY:
Inclusion Criteria:

* Age >50 years old
* Diagnosed with type 2 diabetes
* HbA1c >64mmol/mol

Exclusion Criteria:

1. (History of) malignant diseases or any clinically significant medical condition that could interfere with the conduct of the study in the opinion of the investigator.
2. Chronic or recent infections and/or clinical signs of infection and/or a plasma C-reactive protein above 10ng/ml
3. Auto-immune diseases (including type 1 diabetes)
4. Recent or chronic immunosuppressant or antibiotic usage
5. Use of any GLP1R-agonist at baseline or prior intolerance to use of GLP1R-agonists.
6. Inability or unwillingness to comply with the protocol requirements, or deemed by investigator to be unfit for the study.
7. Uncontrolled hypertension (systolic blood pressure > 180mmHg, diastolic blood pressure > 100mmHg)
8. Uncontrolled chronic inflammatory conditions, including gout.
9. Women of childbearing age who are not using effective contraceptives.
10. Heart failure New York Heart Association (NYHA) class IV at screening visit.
11. Active liver disease or hepatic dysfunction, defined as aspartate aminotransferase (ASAT) or alanine aminotransferase (ALAT) ≥ 2 times the upper limit of normal (ULN) at screening visit.
12. Pancreatitis in medical history.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Difference in coronary 68Ga-Dotatate uptake after treatment. | 6 months
  The within subject comparison of 68Ga-Dotatate uptake in the coronary arteries before and after semaglutide treatment, expressed as a difference in TBRmax.

SECONDARY OUTCOMES:
Difference in bone marrow aspirates after treatment. | 6 months
  The within subject comparison of bone marrow aspirates before and after semaglutide treatment, expressed as a difference in stem cell count.

CONTACTS AND LOCATIONS:
Locations (1):
- AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No